CLINICAL TRIAL: NCT02237157
Title: A Dose Escalation Safety Study of Locally-Delivered (Intra-Arterial) Gemcitabine in Unresectable Adenocarcinoma of the Pancreas
Brief Title: A Dose Escalation Safety Study of Locally-Delivered Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RenovoRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RR1
Record Dates: First submitted 2014-09-08; First posted 2014-09-11 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; unresectable; gemcitabine; device; local delivery; chemoembolization
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: Subjects receive a gradual increase of drug dose, until the full systemic dose is administered. Cycle 1: 250mg/m2. Cycle 2: 500mg/m2. Cycle 3: 750mg/m2. Cycle 4: 1000mg/m2.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Gemcitabine, Local Delivery (Dose 1) (Other): Gemcitabine; 1 cycle, two doses per cycle; 250mg/m2 dose
  Interventions: Drug: Gemcitabine, local delivery
- Gemcitabine, Local Delivery (Dose 2) (Other): Gemcitabine; 1 cycle, two doses per cycle; 500mg/m2 dose
  Interventions: Drug: Gemcitabine, local delivery
- Gemcitabine, Local Delivery (Dose 3) (Other): Gemcitabine; 1 cycle, two doses per cycle; 750mg/m2 dose
  Interventions: Drug: Gemcitabine, local delivery
- Gemcitabine, Local Delivery (Dose 4) (Other): Gemcitabine; 1 cycle, two doses per cycle; 1000mg/m2 dose
  Interventions: Drug: Gemcitabine, local delivery

INTERVENTIONS:
Drug: Gemcitabine, local delivery — Intra-arterial targeted drug delivery
  Other Names: Gemzar

SUMMARY:
A dose escalation, safety study of local (intra-arterially) delivered gemcitabine to the pancreas using the RenovoCath R120 catheter to determine the maximum tolerated dose.

DETAILED DESCRIPTION:
Patients diagnosed with unresectable pancreatic cancer who may or may not have had prior chemotherapy or radiation therapy may be eligible to enroll in this dose escalation study to determine the maximum tolerated dose of gemcitabine to be delivered locally to the pancreatic tumors using the RenovoCath R120 catheter. Patients enrolled may receive up to 8 catheterizations for delivering gemcitabine directly to the pancreatic tumors starting at a reduced dose( 1/4 of standard i.v. gemcitabine dose), then every two doses, increase the dose by 25% if there are no toxicities up to a maximum dose of 1000 mg/m2. There are four cycles, with two doses per cycle. Imaging studies will be conducted as well as assessment for standard, myelosuppresive and gastric toxicities will be assessed. Pain will also be measured throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if all of the following criteria are met:

1. Males and female subjects 18 years of age and older.
2. Subjects with locally advanced unresectable adenocarcinoma (cytological or histologic proof required) of the pancreas.. Patients with islet cell tumors are not eligible.
3. No clinical evidence of distant metastases, excluding single liver metastasis and local lymph node involvement. Patients with more than a single liver metastasis and/or other metastases who have already failed systemic chemotherapy and/or are on a break from systemic chemotherapy who are not surgical candidates can also qualify for this study.
4. Karnofsky Performance Status (KPS) >60.
5. Adequate renal, and bone marrow function described as:

   1. Leukocytes ≥ 3,000/uL
   2. Absolute neutrophil count ≥ 1,500/uL
   3. Platelets ≥100,000/uL
   4. Serum creatinine ≥2.0 mg/dL. Creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than 40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula.
   5. Hemoglobin ≥8.5 g/dL (may be receiving supportive therapy)
   6. PT/PTT (WNL)
6. Adequate Hepatic function (endoscopic or percutaneous drainage as needed) described as:

   1. Total bilirubin ≤3 times UNL (less than or equal to 2 mg/dL)
   2. AST (SGOT)/ALT (SGPT) ≤ 5 times ULN or ≤5 times ULN in the setting of liver metastases.
   3. Lipase and Amylase within normal limits.
7. Capable of understanding the purpose and risks of the study and willing to provide written informed consent and to comply with the procedures

Exclusion Criteria:

Subjects will be excluded from participation in the study if any of the following criteria are met:

1. Have a known sensitivity to gemcitabine.
2. Identification of metastatic disease, with the exception of single liver metastases or local lymph node involvement. Patients with more than a single liver metastasis and/or other metastases who have already failed systemic chemotherapy and/or are on a break from systemic chemotherapy who are not surgical candidates can also qualify for this study.
3. Evidence of coagulopathy.
4. Inability or unwillingness to comply with study procedures and/or follow-up procedures.
5. Evidence of infection or other coexisting medical condition, which in the opinion of the investigator would preclude administration of gemcitabine.
6. Patients with uncontrolled congestive heart failure, unstable angina and myocardial infarction within 3 months.
7. Female patient who is pregnant, nursing or planning on becoming pregnant.
8. Current enrollment and participation in another clinical study or prior exposure to an investigational agent within 12 weeks or 5 half-lives (whichever is longer) of anticipated dosing on Day 1 of this study.
9. Have known brain metastases.
10. Have had any major surgery within four weeks of enrollment.
11. Have any clinically detectable ascites.
12. Have uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
13. Have serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
14. Other invasive malignancies within the past 3 years (with the exception of non-melanoma skin cancers, non-invasive bladder cancer or prostate cancer) not approved by the Medical Monitor (contact MM in event of prior diagnosis with malignancy to discuss enrollment status).
15. Have had any chemotherapy or systemic corticosteroids within 2 weeks of study entry.
16. Have acquired, hereditary or congenital immunodeficiency's including cellular immunodeficiencies, hypogammaglobulinemia and dysgammaglobulinemia or hepatitis.
17. Have a prior history of a documented hemolytic event.
18. Is HIV-positive or Hepatitis positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiali Li, MD, Principal Investigator — El Camino Hospital
Locations (2):
- United States (2):
  - El Camino Hospital, Oncology, Mountain View, California
  - Florida Hospital, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hatoum H, Rosemurgy A 2nd, Bastidas JA, Zervos E, Muscarella P 2nd, Edil BH, Cynamon J, Johnson DT, Thomas C, Swinson BM, Nordgren A, Vitulli P, Nutting C, Gipson M, Tsobanoudis A, Agah R. Treatment of locally advanced pancreatic cancer using localized trans-arterial micro perfusion of gemcitabine: combined analysis of RR1 and RR2. Oncologist. 2024 Aug 5;29(8):690-698. doi: 10.1093/oncolo/oyae178. PMID 39049803

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who complete a cycle ("arm"/"period") then proceed to receive the next higher dose.
Groups:
- Gemcitabine, Local Delivery (Dose 1): Gemcitabine; 1 cycles, two doses per cycle; 250mg/m2 dose
  Gemcitabine, local delivery: Intra-arterial targeted drug delivery
- Gemcitabine, Local Delivery (Dose 2): Gemcitabine; 1 cycles, two doses per cycle; 500mg/m2 dose
  Gemcitabine, local delivery: Intra-arterial targeted drug delivery
- Gemcitabine, Local Delivery (Dose 3): Gemcitabine; 1 cycles, two doses per cycle; 750mg/m2 dose
  Gemcitabine, local delivery: Intra-arterial targeted drug delivery
- Gemcitabine, Local Delivery (Dose 4): Gemcitabine; 1 cycles, two doses per cycle; 1000mg/m2 dose
  Gemcitabine, local delivery: Intra-arterial targeted drug delivery
Period: Gemcitabine, Local Delivery (Dose 1)
Arm/Group | Gemcitabine, Local Delivery (Dose 1) | Gemcitabine, Local Delivery (Dose 2) | Gemcitabine, Local Delivery (Dose 3) | Gemcitabine, Local Delivery (Dose 4)
Started | 20 | 0 | 0 | 0
Completed | 16 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Gemcitabine, Local Delivery (Dose 2)
Arm/Group | Gemcitabine, Local Delivery (Dose 1) | Gemcitabine, Local Delivery (Dose 2) | Gemcitabine, Local Delivery (Dose 3) | Gemcitabine, Local Delivery (Dose 4)
Started | 0 | 15 | 0 | 0
Completed | 0 | 15 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Gemcitabine, Local Delivery (Dose 3)
Arm/Group | Gemcitabine, Local Delivery (Dose 1) | Gemcitabine, Local Delivery (Dose 2) | Gemcitabine, Local Delivery (Dose 3) | Gemcitabine, Local Delivery (Dose 4)
Started | 0 | 0 | 11 | 0
Completed | 0 | 0 | 11 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Gemcitabine, Local Delivery (Dose 4)
Arm/Group | Gemcitabine, Local Delivery (Dose 1) | Gemcitabine, Local Delivery (Dose 2) | Gemcitabine, Local Delivery (Dose 3) | Gemcitabine, Local Delivery (Dose 4)
Started | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine, Local Delivery: Gemcitabine; 4 cycles, two doses per cycle; dose escalation
  Gemcitabine, local delivery: Intra-arterial targeted drug delivery
Arm/Group | Gemcitabine, Local Delivery
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Median (Standard Deviation); unit: years] | 67.5 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated Dose of Gemcitabine to be Delivered Locally to the Pancreas
Description: Maximum Tolerated Dose (MTD) of gemcitabine administered intra-arterially to the pancreatic tumor(s) using the RenovoCath™ RC120 catheter.
  One week post treatment, toxicities will be assessed to determine if there is a pre-defined Dose Limiting Toxicity necessitating dose stopping or holding.
Time Frame: 1 week post treatment
Measure: Number; unit: mg/m^2
Arm/Group | Gemcitabine, Local Delivery
Number analyzed (Participants) | 20
mg/m^2 | 1000

2. Secondary Outcome: CA19-9 Tumor Reduction
Description: Measurements of CA19-9 tumor marker are measured pre-treatment and at various time points (starting with one week) post treatment.
Time Frame: 1 week after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment period, an average of 2.5 months
Arm/Group | Gemcitabine, Local Delivery (Dose 1) | Gemcitabine, Local Delivery (Dose 2) | Gemcitabine, Local Delivery (Dose 3) | Gemcitabine, Local Delivery (Dose 4)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/15 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 5/20 | 4/15 | 3/11 | 2/8
Other Adverse Events (participants affected / at risk) | 7/20 | 7/15 | 4/11 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Local Delivery (Dose 1) (N=20) | Gemcitabine, Local Delivery (Dose 2) (N=15) | Gemcitabine, Local Delivery (Dose 3) (N=11) | Gemcitabine, Local Delivery (Dose 4) (N=8)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal Obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative Arterial Injury / Dissection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Intraoperative Arterial Injury - Lower Extremity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Abdominal (NOS) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Local Delivery (Dose 1) (N=20) | Gemcitabine, Local Delivery (Dose 2) (N=15) | Gemcitabine, Local Delivery (Dose 3) (N=11) | Gemcitabine, Local Delivery (Dose 4) (N=8)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative arterial injury - lower extremity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative arterial injury - pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Median arcuate ligament syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No